CLINICAL TRIAL: NCT00646633
Title: Improving Fatigue: A Pilot Study of Acupuncture and Patient Education for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 06-08-010
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2008-03

CONDITIONS: Fatigue
Keywords: Cancer; Acupuncture
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Acupuncture Therapy; Patient Education as Topic; Medicine, Chinese Traditional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture & educ (Active Comparator): Patients will receive a total of 8 acupuncture treatments. In each of the first four sessions, they will also receive patient education.
  Interventions: Procedure: Acupuncture and patient education
- 2. Standard care (No Intervention): Patients in the control arm will continue to receive standard care from their physician.

INTERVENTIONS:
Procedure: Acupuncture and patient education — Acupuncture involves the insertion of extremely thin needles, much thinner than those used for drawing blood, into very specific acupuncture points. Patients will receive a total of 8 acupuncture treatments, each lasting 50 minutes. Patient education will be delivered to individuals over the course of approximately 50 minutes for each of the four sessions; topics will include acupressure, nutrition, exercise, stress management, and lifestyle advice.
  Other Names: Traditional Chinese Medicine, Integrative East-West Medicine
  Arms: Acupuncture & educ

SUMMARY:
Based on the investigators clinical experience in patients with chronic disease (Hui, Hui, and Johnston, 2006; Hays et al 2005), a review of the literature (Johnston, Xiao and Hui 2007), and inspired by Vickers and colleagues (PMID: 15117996), the investigators carry out a pilot study that investigates if acupuncture combined with patient education will relieve fatigue in patients who have completed primary treatment for breast cancer.

DETAILED DESCRIPTION:
Patients will be randomly assigned to one of the two groups. Our hypothesis is that patients in the acupuncture/education group will experience greater relief of fatigue than those in the standard care group.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 65 years of age
2. Patient has a rounded Brief Fatigue Inventory score of 4 or greater
3. Patient is in a stable clinical condition

Exclusion Criteria:

1. Severe anemia (hemoglobin level less than 9 g/dL, hematocrit level less than 30, decline in hemoglobin of 2 g/dL in the previous month, or active treatment for anemia)
2. Karnofsky Performance Status below 70
3. Acupuncture treatment in the previous 6 months
4. Fatigue before cancer diagnosis
5. Patient is mentally incapacitated or unfit to provide informed consent or participate in an interview
6. Patient has the potential for serious bleeding due to inherited diseases such as hemophilia
7. Patient is taking medications that are either fatigue-inducing or have sedating properties
8. Patient is unavailable by telephone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Fatigue as measured by the Brief Fatigue Inventory | prior to beginning of treatment and after treatment ends. Up to an average of 44 weeks.

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQoL) as measured by the SF36 | prior to beginning of treatment and after end of treatment. Up to an average of 44 weeks.
Pain as measured by an analog scale | prior to beginning of treatment and after conclusion of treatment. Up to an average of 44 weeks.
Cognitive complaints as measured by the FACT-COG | prior to the beginning of treatment and after end of treatment. Up to an average of 44 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Kit Hui, M.D., Principal Investigator — UCLA Center for East-West Medicine, 1033 Gayley Ave, Suite 111, Los Angeles, CA 90024
Locations (1):
- UCLA Center for East-West Medicine, Santa Monica, California, United States

REFERENCES:
- [Background] Hui KK, Hui EK, Johnston MF. The potential of a person-centered approach in caring for patients with cancer: a perspective from the UCLA center for East-West medicine. Integr Cancer Ther. 2006 Mar;5(1):56-62. doi: 10.1177/1534735405286109. PMID 16484714
- [Background] Hays RD, Brodsky M, Johnston MF, Spritzer KL, Hui KK. Evaluating the statistical significance of health-related quality-of-life change in individual patients. Eval Health Prof. 2005 Jun;28(2):160-71. doi: 10.1177/0163278705275339. PMID 15851771
- [Background] Johnston MF, Xiao B, Hui KK. Acupuncture and fatigue: current basis for shared communication between breast cancer survivors and providers. J Cancer Surviv. 2007 Dec;1(4):306-12. doi: 10.1007/s11764-007-0035-9. Epub 2007 Oct 31. PMID 18648966
- [Background] Vickers AJ, Straus DJ, Fearon B, Cassileth BR. Acupuncture for postchemotherapy fatigue: a phase II study. J Clin Oncol. 2004 May 1;22(9):1731-5. doi: 10.1200/JCO.2004.04.102. PMID 15117996
- [Derived] Johnston MF, Hays RD, Subramanian SK, Elashoff RM, Axe EK, Li JJ, Kim I, Vargas RB, Lee J, Yang L, Hui KK. Patient education integrated with acupuncture for relief of cancer-related fatigue randomized controlled feasibility study. BMC Complement Altern Med. 2011 Jun 25;11:49. doi: 10.1186/1472-6882-11-49. PMID 21703001